CLINICAL TRIAL: NCT05554614
Title: Behind the Wheel (BTW) Smartphone Application: Utilizing Technology to Quantify Driving Behaviors
Brief Title: Behind the Wheel (BTW) Smartphone Application
Acronym: BTW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Motao Zhu (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Motao Zhu, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00002565; FP00001219 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2022-07-13; First posted 2022-09-26 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: High-risk Driving Events

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- BTW app with reward-based feedback (Experimental): Teens will install the BTW app with reward-based feedback. This tracks driving performance while providing individualized driving feedback using gamification concepts.
  Interventions: Behavioral: BTW app with reward-based feedback; Behavioral: BTW app with situational supervised driving practice
- BTW app with situational supervised driving practice (Experimental): Teens will install the BTW app the same as the app with reward-based feedback in conjunction with a situational supervised driving practice intervention for teen-parent dyads.
  Interventions: Behavioral: BTW app with situational supervised driving practice
- Sham BTW app (Sham Comparator): Teens will install the sham BTW app with driving performance tracking only.
  Interventions: Behavioral: Sham BTW app

INTERVENTIONS:
Behavioral: BTW app with reward-based feedback — Teen drivers will be notified of their weekly driving performance via a driving safety score with information on the types of high-risk driving behaviors committed as well as progress on maintaining and/or improving weekly safe driving behaviors. Educational materials on different driving situations and scenarios associated with the high-risk driving behaviors (e.g. 90-second videos) will be provided for the driver to review at any point and time. Information on these driving behaviors and the education material will be provided via push notifications from the BTW app. Weekly leader boards will show the driver's driving safety score in comparison to other drivers of the same age. Consistently high driver safety scores in certain driving skill areas (e.g., cornering) and a total overall score above 70% of other users on that skill or total score will unlock gamification-based rewards (e.g., driving safety badges, driving safety score leader board, group challenges with winners).
  Arms: BTW app with reward-based feedback
Behavioral: BTW app with situational supervised driving practice — Teen drivers will be provided bi-weekly push-notifications from the BTW app notifying them of situational supervised driving practice activities that are to be completed during the assigned week. There are 12 situational supervised driving activities and six skill-building driving activities (Table 1). Skill-building sessions are assigned for off weeks during the first half of the six months (weeks 2-12), allowing for skills to be further developed when the situations are encountered for a second time (weeks 15-23). Parents will be prompted to directly log situational supervised and skill-building driving activities in the app after the session within the BTW app to obtain the module completion date and duration time.
  Arms: BTW app with reward-based feedback; BTW app with situational supervised driving practice
Behavioral: Sham BTW app — Teens will be provided links to passive education materials and information on car maintenance every week. They will not be given feedback on their driving performances.
  Arms: Sham BTW app

SUMMARY:
The purpose of this study is to find out if a phone app can help the learning-to-drive process among teenagers and novice drivers.

DETAILED DESCRIPTION:
This project will assess the feasibility and preliminary efficacy of an app (BTW) to quantify driving behaviors and promote safe driving in adolescents who are beginning their learner period of licensure. 90 teens and their corresponding parents/guardians will be randomized into one of three study groups. Researchers aim to test the feasibility of the BTW app on acceptance and retention, evaluate the preliminary efficacy of the BTW app with a teen-parent dyad intervention on driving performance after using the BTW app for six months, and investigate the long-term effects of the BTW app intervention on driving performance and safety attitudes among teens.

ELIGIBILITY:
Inclusion criteria:

* Teen participants must be between the ages of 15.5-17 years old at the time of enrollment
* Participants must have one parent and/or legal guardian who agrees to participate in the study.
* Participants' parents must possess car insurance with at least state-minimum coverage.
* Participants must be willing to fulfill the minimum requirements of the Ohio GDL system.
* Driver must complete a driver education class at a licensed driver training school with 24 hours of classroom or online instruction and 8 hours of driving time; driver must complete 50 hours of driving with at least 10 hours of night driving; driver must hold the permit for at least 6 months.
* Participants must have a functioning smartphone and active smartphone account compatible for the BTW app.
* To prevent any interference from another driving-related study, participants must agree not to enroll in other driving-related research/driving performance app during the study period.
* Participants must be willing to be randomized and comply with study requirements.
* Participants must speak and read English.
* Participants must be a US citizen or have permanent resident status.

Exclusion criteria:

- Drivers younger than 15.5 will be excluded because Ohio does not issue a temporary instruction driving permit identification card (i.e., learner's driving permit) starting the GDL process until age 15.5.

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2023-02-19 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
High-risk driving events | Baseline to 6 months post randomization
  Number of high-risk driving events (harsh breaking, accelerating, and cornering events) per 1,000 miles driven. Higher numbers signify more high-risk driving events.

SECONDARY OUTCOMES:
Speeding and near-crash events | Baseline to 6 months post randomization
  Instances of speeding and number of near crashes and crashes per 1,000 miles driven. Higher numbers signify more near-crash events.

OTHER OUTCOMES:
Self-reported high risk driving behaviors | 18-month study period
  Self-reported frequency of high risk driving behaviors including speeding, distracted driving and driving under the influence of alcohol or drugs.
Self-reported driving safety attitudes | 18-month study period
  The distribution of attitudes towards traffic safety behaviors, including speeding, distracted driving, and driving under the influence of alcohol or drugs, measured through self-report on 4-point Likert scales.
Self-reported traffic violations | 18-month study period
  The number of traffic violations, including speeding, intoxicated driving, and distracted driving, measured through self-report on a questionnaire.
Police-reported traffic violations | 18-month study period
  Number of police-reported crashes and traffic violations. Higher numbers signify more crashes and violations.

CONTACTS AND LOCATIONS:
Overall Officials: Motao Zhu, MD, MS, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No